CLINICAL TRIAL: NCT04739956
Title: Psychological Impact of Pregnancy of Unknown Location
Acronym: SOUL
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19QC5631
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy of Unknown Location; Ectopic Pregnancy; Anxiety
Keywords: Pregnancy of unknown location; PUL; Ectopic pregnancy; Anxiety
MeSH Terms: conditions — Pregnancy, Ectopic; Anxiety Disorders | interventions — Point-of-Care Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: point of care (POC) result not shared: Patients in this phase of the study will not be provided with the POC BhCG result. They will await the laboratory result. Simultaneously we will ascertain reliability of POC in clinical practice during this time.
  Interventions: Other: The Hospital and Anxiety Depression Scale; Other: Point of care testing (POCT)
- Patient: point of care (POC) result shared: Patients in this phase will be informed of the POC test result, which will reduce the time to which they receive the result. Prior to transfer to this phase, correlation between POC and laboratory BhCG levels will be calculated in order to confirm its reliability by creating a correlation curve using the data.
  Interventions: Other: The Hospital and Anxiety Depression Scale; Other: Point of care testing (POCT)

INTERVENTIONS:
Other: The Hospital and Anxiety Depression Scale — Patients and partners will be asked to complete the questionnaire at three time points: 1) On classification of PUL at time zero once blood is taken, 2) at the 48-hour time point after blood is taken (if 48 hour bloods are required for the patient); and 3) after definitive diagnosis and management.
Other: Point of care testing (POCT) — Patients will have 1ml sample of blood taken for POCT at two time points: 1) On classification of PUL at time zero at the same time as when routine blood samples taken; and 2) at the 48-hour time point at the same time as when routine blood samples are taken (if 48 hour bloods are required).

SUMMARY:
To assess the psychological impact of pregnancy of unknown location (PUL) classification pending a final diagnosis.

DETAILED DESCRIPTION:
PUL is a syndrome of early pregnancy composed of a positive urine pregnancy test without the visualisation of a pregnancy on trans-vaginal ultrasound (TVUS). The current method for risk stratifying a PUL is via serum BhCG levels at the time of identification of PUL and after 48 hours, in order to ascertain the viability of the pregnancy. Patients and their partners need to wait for this result before a management plan can be adopted, taking at least 2-3 hours. There is a clear need for the patient care pathway to evolve in order to aid and improve the management of women classified with a PUL. By using point-of-care BhCG testing, the investigators hope to shorten the time to management. The investigators therefore propose that shortening the time interval would reduce psychological morbidity. This is a prospective cohort observational study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending the Early Pregnancy Unit in the first trimester (up to 14 weeks gestation) with a pregnancy of unknown who are over 18 years old and are able to give consent.

Exclusion Criteria:

* Presence diagnosed with cancer
* The presence of an acute medical condition
* Patients/partners aged less than 18 years
* Patients or partners who cannot give fully informed study consent (language or learning impairment)
* Presence of a viable intrauterine pregnancy, ectopic pregnancy and miscarriage.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women attending the Early Pregnancy Unit in the first trimester (up to 14 weeks gestation) with a pregnancy of unknown who are over 18 years old and are able to give consent.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kyriacou C, Yang W, Kapur S, Maheetharan S, Pikovsky M, Parker N, Barcroft J, Bobdiwala S, Sur S, Stalder C, Gould D, Ofili-Yebovi D, Day A, Unsworth N, Wilkes EH, Tan T, Bourne T. Ambulatory human chorionic gonadotrophin (hCG) testing: a verification of two hCG point of care devices. Clin Chem Lab Med. 2023 Oct 30;62(4):664-673. doi: 10.1515/cclm-2023-0703. Print 2024 Mar 25. PMID 37886834

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient: Point of Care (POC) Result Not Shared | Patient: Point of Care (POC) Result Shared
Started | 74 | 76
Completed | 73 | 75
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient: Point of Care (POC) Result Not Shared | Patient: Point of Care (POC) Result Shared | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (5.1) | 34 (6) | 34 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 76 | 150
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 44 | 91
  Black | 6 | 8 | 14
  Asian | 11 | 14 | 25
  Mixed | 0 | 3 | 3
  Other | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 74 | 76 | 150

OUTCOME MEASURES:

1. Primary Outcome: Psychological Morbidity
Description: Psychological morbidity will be assessed using the Hospital Anxiety and Depression Scale on time of PUL classification, 48 hours from PUL classification and following final diagnosis and management. For both Anxiety and Depression, participants can score anywhere from 0 to 21. Score of 11 and above indicate moderate to severe anxiety and depression.
Time Frame: 0 hours, 48 hours and point of diagnosis (within 2 wees)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient: Point of Care (POC) Result Not Shared | Patient: Point of Care (POC) Result Shared
Number analyzed (Participants) | 73 | 75
score on a scale
  0hrs anxiety score | 10 (5) | 10 (4)
  0hrs depression score | 5 (4) | 5 (4)
  48hrs anxiety score | 10 (5) | 9 (4)
  48hrs depression score | 6 (4) | 5 (4)

ADVERSE EVENTS:
Time Frame: 15 months
Description: Serious and other [non-serious] adverse events were not observed on blood sample collection. The rest of the study was with quesionnaires only: there was no expectation of exposure to any risks after blood sample collection, as the remaining of the study involved only the completion of quesionnaires by the patients.
Groups:
- Patient: Point of Care (POC) Result Not Shared; Patient: Point of Care (POC) Result Shared: Serious and other [non-serious] adverse events were not collected or assessed as part of the study.
Arm/Group | Patient: Point of Care (POC) Result Not Shared | Patient: Point of Care (POC) Result Shared
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/76
Other Adverse Events (participants affected / at risk) | 0/74 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT04739956/Prot_SAP_000.pdf